CLINICAL TRIAL: NCT07366398
Title: Hyaluronic Acid as Adjunctive to Chlorhexidine Mouthwash for Gingivitis: RCT
Brief Title: Hyaluronic Acid Mouthwash as Adjunct
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, PI, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACU-Per2
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Gingivitis; Chronic
MeSH Terms: conditions — Gingivitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine mouthwash (Active Comparator)
  Interventions: Drug: Chlorhexidine 0,12%
- Hyaluronic acid + Chlorhexidine mouthwash (Active Comparator)
  Interventions: Drug: Hyaluoric acid mouthwash; Drug: Chlorhexidine 0,12%

INTERVENTIONS:
Drug: Hyaluoric acid mouthwash — A mouthwash containing both hyaluronic acid
  Arms: Hyaluronic acid + Chlorhexidine mouthwash
Drug: Chlorhexidine 0,12% — mouthwash of chlorhexidine 0.12%

SUMMARY:
Patients were instructed to use 2 different mouthwashes after performing professional tooth cleaning. The effect of each of the 2 mouthwashes was detected.

DETAILED DESCRIPTION:
The study tests the efficacy of hyaluronic acid (HYL) mouthwash as adjunct to Chlorhexidine (CHX) mouthwash compared to Chlorhexidine mouthwash only in 16 gingivitis patients. Patients were randomly assigned to either control group received (Chlorhexidine mouthwash) or test group received (hyaluronic acid + Chlorhexidine mouthwash). Clinical parameters and patient reported outcomes as post-operative questionnaire were assessed at baseline and seven days post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with gingivitis

Exclusion Criteria:

* pregnant or lactating females and current smokers

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 7 days
  % of gingival sites where bleeding occurred on periodontal probing is registered out of total gingival sites

SECONDARY OUTCOMES:
Plaque index | 7 days
  % of gingival sites where plaque accumulates is registered out of total gingival sites
Patient's satisfaction questionnaire | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ahram Canadian University, Giza, Egypt